CLINICAL TRIAL: NCT06198153
Title: Comparative Effects of Stationary Cycling and Progressive Functional Training on Balance and Motor Control of Lower Extremity in Children With Cerebral Palsy
Brief Title: Effects of Stationary Cycling and Progressive Functional Training in Cerebral Palsy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0751
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy
Keywords: : Balance, Cerebral palsy, Cycling,; Motor control; Functional training,
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stationary Cycling (Active Comparator): This group will receive stationary cycling for 6 weeks.
  Interventions: Other: Stationary Cycling
- Progressive Functional Training (Experimental): This group will receive Progressive Functional Training programs for 6 weeks.
  Interventions: Other: Progressive Functional Training

INTERVENTIONS:
Other: Stationary Cycling — In addition to the conventional physical therapy, children in this group will receive 10-15 minutes of stationary cycle training, 3 times a week for 6 weeks.
  Arms: Stationary Cycling
Other: Progressive Functional Training — In addition to the conventional physical therapy, the training will follow a 6-week progressive functional training program for lower extremities. These exercises will include sit-to-stand exercise, lateral/forward step-up exercise (i.e. climbing a stair or stepping up onto a kerb), and half-knee rise exercise (i.e. rising from the ground). All exercises will be performed in 1-3 sets of 10-15 repetitions, with a 90 second rest in between the sets. Each exercise will be performed within 10-15 minutes. Training session will be given 3 times a week. During the training, intensity will be progressively increased by increasing the repetitions
  Arms: Progressive Functional Training

SUMMARY:
Cerebral palsy is not a progressive disease but movement problem and musculoskeletal disorders in cerebral palsy change with time. Children with CP usually with the lower limb involvement presents with muscle weakness, limited muscular control which results in muscular insufficiency, coordination and balance impairment. These impairments effect the normal activities of child in daily living. There are many children who have good cognition but poor lower limb coordination which is leading cause of disability in them and multiple factors are responsible for them like lake of awareness in parents, no time, expensive therapy program and inappropriate techniques.

DETAILED DESCRIPTION:
The study will be randomized clinical trial and will be conducted in Bahawalpur. The study will be completed in time duration of 6 months after approval of synopsis. Non probability convenience sampling technique will be used and 22 children will be recruited in the study meeting the inclusion criteria. The participants will be divided into two groups through randomization using lottery method. Group A will perform 10-15 minutes of stationary cycle training, 3 times a week for 6 weeks. While group B will be given progressive functional training 3 times a week for 10-15 minutes for 6 weeks. Pediatrics balance scale will be used to measure functional balance skills and GMFS scale will be used to measure gross motor function. The data will be assessed at the baseline and after 6 weeks of intervention. After data collection data will be analyzed by using SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* • Children with cerebral palsy (Hemiplegic)

  * Age: 4 to 10 years
  * Able to sit without foot or arm support
  * Children with level I & II on Gross motor function classification system
  * Normal cognitive function; can understand and follow command

Exclusion Criteria:

* • Children with mental retardation.

  * Visual and auditory disorders.
  * History of any surgical procedure.
  * Any infections, unstable seizures, etc.
  * Fixed deformities or contractures of lower limbs.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
GMFM Scale | 6weeks
  The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy. The scoring key is meant to be a general guideline. (13) However, most of the items have specific descriptors for each score. It is imperative that the guidelines contained in the manual be used for scoring each item.
  Scoring Key:
  0= does not initiate
  1. initiates
  2. partially completes
  3. completes 9 (or leave blank) = not tested (NT) [used for the GMAE-2 scoring*] It is important to differentiate a true score of -0‖ (child does not initiate) from an item which is Not Tested (NT) if you are interested in using the GMFM-66 Ability Estimator (GMAE) Software. It is reliable with 95% confidence interval=0.965-0.994. The validity with 95% confidence interval=0.972-0.997
Pediatrics Balance Scale | 6 weeks
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children. (15) The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points Reliability testing performed with a sample of 20 children ages 5-15 years old with mild to moderate motor impairments showed good test-retest reliability (ICC=0.998) and good interrater reliability (ICC=0.997).

CONTACTS AND LOCATIONS:
Overall Officials: Aneeza Maryam, MS*, Principal Investigator — Riphah International University
Locations (1):
- Imran Amjad, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ansa OEO, Mprah KW, Moses MO, Owusu I, Acheampong E. Effect of Community-Based Functional Aerobic Training on Motor Performance and Quality of Life of Children with Spastic Cerebral Palsy. Ethiop J Health Sci. 2021 Mar;31(2):381-392. doi: 10.4314/ejhs.v31i2.21. PMID 34158790